CLINICAL TRIAL: NCT05958004
Title: Application Value of Biopsy Free Technique for Prostate Specific Antigen Grey Area Prostate Cancer Based on 18F-Prostate Specific Membrane Antigen-1007 Positron Emission Tomography/Computerized Tomography
Brief Title: The Application Value of Prostate Specific Membrane Antigen PET/CT in Biopsy Free of PSA Grey Area Prostate Cancer
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-367
Record Dates: First submitted 2023-07-06; First posted 2023-07-24 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Prostatic Neoplasms
Keywords: PET/CT; PSMA; PSA grey area
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — RNA expression and gene mutation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Prostate Cancer: Participants who are suspected of prostate cancer due to elevated PSA but have not received any treatment and eventually confirmed non-prostate cancer after biopsies
- Prostate Cancer: Participants who are suspected of prostate cancer due to elevated PSA but have not received any treatment and eventually confirmed prostate cancer after biopsies

SUMMARY:
The goal of this observational study is to establish an evaluation system for accurate identification of prostate cancer and clinical significant prostate cancer in patients in the PSA gray zone. The main questions it aims to answer are: proportion of men who could have avoided biopsy with positive PSMA-PET and no clinically significant cancer detected on biopsy.

Participants will: 1. undergo PSMA PET/CT and multiparametric MRI; and 2. undergo prostate biopsy

Researchers will compare the diagnostic performance of PSMA PET/CT and multiparametric MRI for prostate cancer and clinical significant prostate cancer to see if there are differences.

DETAILED DESCRIPTION:
Prostate Specific Antigen (PSA) is a serine protease secreted by prostate epithelial cells, which is a tumor marker of prostate cancer. At present, PSA<4 ng/ml is considered as the normal value, and PSA 4-10 ng/ml is considered as the gray value. PSA>10 ng/ml should be highly suspected of prostate cancer. Prostate biopsy is still the gold standard for the diagnosis of prostate cancer. However, as an invasive procedure, it can cause many complications such as pain, bleeding, lower urinary tract symptoms and infection. There is a growing trend to reduce unnecessary prostate biopsies.

Prostate specific membrane antigen (PSMA) is a membrane-bound enzyme that is highly expressed in more than 90% of prostate cancer lesions and has become an important target for molecular imaging of prostate cancer. In recent years, radioactive nuclide 18F labeling targeting PSMA positron emission tomography/computed tomography (PET/CT) has shown important clinical application value in prostate cancer recurrence monitoring.

The goal of this observational study is to establish an evaluation system for accurate identification of prostate cancer and clinical significant prostate cancer in patients in the PSA gray zone.

Participants will: 1. undergo PSMA PET/CT and multiparametric MRI; and 2. undergo biopsy

Researchers will compare the diagnostic performance of PSMA PET/CT and multiparametric MRI for prostate cancer and clinical significant prostate cancer to see if there are differences.

ELIGIBILITY:
Inclusion Criteria:

* PSA (4-10 ng/mL)
* MRI and PSMA PET/CT were not contraindicated
* Did not receive prostate-related treatment
* There are no contraindications to biopsy

Exclusion Criteria:

* Coexisting with other malignancies

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -Patients with elevated PSA levels in the First Affiliated Hospital of Xi'an Jiaotong University be included in this study with signed informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
detection rate of prostate cancer | about 1 year
  detection rate of prostate cancer
detection rate of clinical significant prostate cancer | about 1 year
  detection rate of clinical significant prostate cancer

SECONDARY OUTCOMES:
gleason score group prediction | about 1 year
  Using biopsy histopathology as standard, patients will be classified as gleason score 6-10. We use PSMA PET and genomics to predict gleason score group
expression level of survival-related genes | about 1 year
  Using RNA sequence to evaluate the expression level of survival-related genes

CONTACTS AND LOCATIONS:
Overall Officials: Zhuonan Wang, Ph.D., Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Luo L, Wang R, Bai L, Shang J, Wang X, Chang R, Dong W, Li Y, Li Y, Liang H, Xie H, Duan X. The accuracy of fluorine 18-labelled prostate-specific membrane antigen PET/CT and MRI for diagnosis of prostate cancer in PSA grey zone. Br J Cancer. 2025 Feb;132(3):253-258. doi: 10.1038/s41416-024-02934-x. Epub 2024 Dec 19. PMID 39702584